CLINICAL TRIAL: NCT04914351
Title: A Phase Ⅰ, Multi-center, Open-label, Single-arm, Dose Escalation, First-in-human Clinical Study of HY-0102 Monotherapy in Patients With Locally Advanced/Metastatic Solid Tumours
Brief Title: HY-0102 Monotherapy in Patients With Locally Advanced/Metastatic Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai HyaMab Biotech Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY-0102-01
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-04

CONDITIONS: Locally Advanced/Metastatic Solid Tumors
Keywords: HY-0102, solid tumors

STUDY DESIGN:
Intervention Model Description: This is a Phase I, first-in-human, single-arm and multi-centre trial to evaluate the safety, tolerability, pharmacokinetics and preliminary antitumor activity of HY-0102 in adult patients with locally advanced/metastatic malignant solid tumors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Cohort 1: 0.03 mg/kg Q2W HY-0102 ivgtt Duration: 26w DLT observation period: 28 days Accelerated dose escalation: One patient will be enrolled. Cohort 2: 0.3 mg/kg Q2W HY-0102 ivgtt Duration: 26w DLT observation period: 28 days Accelerated dose escalation: One patient will be enrolled. Cohort 3: 1 mg/kg Q2W HY-0102 ivgtt Duration: 26w DLT observation period: 28 days Standard 3+3 Dose escalation: Three patients will be enrolled for each dose cohort.
  Cohort 4: 2 mg/kg Q2W HY-0102 ivgtt Duration: 26w DLT observation period: 28 days Standard 3+3 Dose escalation: Three patients will be enrolled for each dose cohort.
  Cohort 5: 4 mg/kg Q2W HY-0102 ivgtt Duration: 26w DLT observation period: 28 days Standard 3+3 Dose escalation: Three patients will be enrolled for each dose cohort.
  Cohort 6: 10 mg/kg Q2W HY-0102 ivgtt Duration: 26w DLT observation period: 28 days Standard 3+3 Dose escalation: Three patients will be enrolled for each dose cohort.
  Interventions: Drug: HY-0102

INTERVENTIONS:
Drug: HY-0102 — Multiple dose cohorts, 60 minute IV infusion, every two weeks, 28 days as a cycle

SUMMARY:
This is a Phase I, first-in-human trial to evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of HY-0102 administered intravenously (IV) once every two weeks in adult patients with locally advanced/metastatic malignant solid tumors.

DETAILED DESCRIPTION:
This is a Phase I, first-in-human trial to evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of HY-0102 administered intravenously (IV) once every two weeks in adult patients with locally advanced/metastatic malignant solid tumors (head and neck, liver, colorectal and lung cancers, etc).

Six dosing cohorts are planned with the dose of 0.03, 0.3, 1, 2, 4 and 10 mg/kg. The first two dose levels (0.03 and 0.3 mg/kg) will each enroll one patient using an accelerated escalation design that will convert to a 3+3 design upon the occurrence of one treatment-related Grade 2 toxicity occurring in the safety evaluation window following the first dose of treatment. After the initial two cohorts are completed, the study will use a standard 3+3 dose escalation design.

The number of enrolled patients is estimated to be up to 32. The dose limiting toxicity evaluation period will be the first 28 days (Cycle 1) and subsequent cycles will be 4 weeks in duration. Patients will receive the investigational drug on Day 1 of cycle 1 followed by 28 days of observation. HY-0102 will be administered IV once every two weeks for Cycle 2 and beyond.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years
2. Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures.
3. Histologically or cytologically confirmed incurable, unresectable, locally advanced or metastatic cancer that is refractory to standard therapies.
4. Prior Therapy

   1. Have progressed on or are intolerant to all standard therapies
   2. Have no available therapies known to confer clinical benefit
5. Measurable or evaluable disease per RECIST v1.1 Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm (≥ 2 cm) by chest x-ray or as ≥10 mm (≥ 1 cm) with CT scan, MRI, or calipers by clinical exam.
6. ECOG performance status 0 or 1; Life expectancy ≥ 3 months.
7. Adequate hepatic function as evidenced by meeting all the following requirements:

   1. Total bilirubin ≤ 1.5 ×within institutional upper limit of normal (ULN); or ≤ 2.5 × institutional ULN for patients who have serum bilirubin increases due to underlying Gilbert's Syndrome or familial benign.
   2. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) ≤ 2.5 × ULN; AST or ALT ≤ 5 × ULN if liver metastases are present.
8. Serum creatinine < 1.5 × ULN and calculated creatinine clearance (CrCL) > 30 mL/min (Cockroft-Gault Equation).
9. Hematological function defined as:

   1. Absolute neutrophil count ≥ 1,500//L without growth factor support in the 2 weeks prior to study entry
   2. Hemoglobin > 9 g/dL without transfusion in the 2 weeks prior to study entry
   3. Platelet count ≥ 75,000/L without transfusion in the 2 weeks prior to study entry
10. Prothrombin time, international normalized ratio or activated partial thromboplastin time < 1.5 × ULN; Use of full dose anticoagulants is permitted. These laboratories should be maintained within the therapeutic range and closely monitored by the Investigator.
11. Recovery, to Grade 0-1, from adverse events related to prior anticancer therapy except alopecia, < Grade 2 sensory neuropathy, lymphopenia, and endocrinopathies controlled with hormone replacement therapy.
12. For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception during study treatment that results in a low failure rate of <1% per year when used consistently and correctly. Female and male patient treated with HY-0102 should continue contraception use for 6 months after the last dose. Such methods include combined (estrogen and progestogen containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion or vasectomized partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.

    * Oral contraception should always be combined with an additional contraceptive method because of a potential interaction with the study drug. The same rules are valid for male patients involved in this clinical trial if they have a partner of childbirth potential. Male patients must always use a condom.
    * Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 7 days prior to initiation of study drug.
    * Women are excluded from birth control if they had had tubal ligation or a hysterectomy.

Exclusion Criteria:

1. Symptomatic central nervous system metastases. Patients with asymptomatic CNS metastases who are radiologically and neurologically stable ≥ 4 weeks following CNS-directed therapy, and are on a stable or decreasing dose of corticosteroids are eligible for study entry.
2. Uncontrolled hypertension (systolic blood pressure >150 mmHg and diastolic blood pressure >90 mmHg), a history of hypertension crisis, or a history of hypertensive encephalopathy.
3. Severe cardiovascular disease, including CVA, TIA, myocardial infarction, or unstable angina within 6 months of study entry; NYHA class III or IV heart failure within 6 months of study entry; Uncontrolled arrhythmia within 6 months of study entry.
4. QTc > 450 ms at baseline; no concomitant medications that would prolong the QT interval; no family history of long QT syndrome [consider QTc < 480 rather than 450]
5. Concurrent malignancy within 5 years prior to entry other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, prostate cancer under active surveillance, prostate cancer that has undergone definitive treatment, ductal carcinoma in situ of the breast, or < T1 urothelial carcinoma.
6. Active infection requiring intravenous therapy within 2 weeks prior to entry.
7. Active HIV, hepatitis B or hepatitis C virus. or

   1. Patients infected with the HIV virus will be eligible if their CD4 count is > 350 cells/mm3 and the patient is on anti-retroviral therapy with an HIV viral load that is below the level of detection.
   2. Active hepatitis B or C. HBV carriers without active disease (HBV DNA titer < 1000 cps/mL or 200 IU/mL), or cured Hepatitis C (negative HCV RNA test) may be enrolled. For patients with hepatocellular carcinoma, patient with chronic infections with hepatitis C virus (treated or untreated); and patients with hepatitis B virus who were treated with antiviral therapy and who had a HBV viral load less than 200 IU/mL may also be enrolled.
8. Active tuberculosis
9. Anticancer therapy or radiation therapy within 5 half-lives or 4 weeks (whichever is shorter) prior to study entry; Palliative radiotherapy to a single area of metastasis is within 2 weeks prior to study entry.
10. Prior treatment with drugs in the same class.
11. Major surgery within 4 weeks prior to study entry; minor surgery within 2 weeks prior to study entry.
12. Allergy to study drug or components of its formulation.
13. No history of a Grade 3-4 allergic reaction to treatment with another monoclonal antibody.
14. Pregnant or breast-feeding females.
15. Women of childbearing potential who do not consent to use two highly effective methods of birth control (including one barrier method) during treatment and for an additional 5 half lives after the last administration of study drug.
16. Men with a partner of childbearing potential who do not consent to use two highly effective methods of birth control (including one barrier method) during treatment and for an additional 5 half lives after the last administration of study drug.
17. Any condition that the investigator or primary physician believes may not be appropriate for participating the study.
18. Live virus vaccine within 30 days prior to study entry.
19. Active autoimmune disease or history of autoimmune disease requiring systemic therapy within 2 years prior to entry except hypothyroidism, vitiligo, Grave's disease, Hashimoto's disease, or Type I diabetes.
20. History of Grade 3-4 immune-related adverse events or immune-related adverse events requiring discontinuation of prior therapies.
21. Use of systemic corticosteroids in a dose equivalent to > 10 mg/d of prednisone or other immunosuppressive agent within 2 weeks prior to entry; Use of inhaled, topical, or ophthalmological steroids are allowed. Short term (< 30 days) uses of corticosteroids at doses equivalent to > 10 mg/d of prednisone (e.g., pre-medication for IV contrast) is allowed.
22. Prior allogeneic stem cell, bone marrow, or solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of Drug Limited Toxicities (DLTs) | From Time of First dose through DLT observation period, 28 days
  To assess by the occurrence of Drug Limited Toxicities (DLTs)
Incidence of Treatment-emergent adverse event (TEAEs) and serious adverse events (SAEs). | From the start of treatment until up to 90 days after the last dose of study drug
  To assess by the occurrence of Treatment-emergent adverse event (TEAEs) and serious adverse events (SAEs)
Number of patients with changes in laboratory parameters from baseline | From the start of treatment until up to 30(±7) days after the last dose of study drug
  To assess safety of HY-0102
Number of patients with changes in electrocariogram (ECG) from baseline | From the start of treatment until up to 30(±7) days after the last dose of study drug
  To assess safety of HY-0102
Number of participants with changes in left ventricular ejection fraction (LVEF) from baseline | From the start of treatment until up to 30(±7) days after the last dose of study drug
  To assess safety of HY-0102
Number of participants with changes in Clinically Significant Vital Sign from baseline | From the start of treatment until up to 30(±7) days after the last dose of study drug
  To assess safety of HY-0102

SECONDARY OUTCOMES:
Cmax (Maximum observed serum concentration) of HY-0102 | From first dose through 30days(±7) days after the last dose of study medication
  Cmax of HY-0102 was observed directly from data
Ctrough (Trough observed serum concentration) of HY-0102 | From first dose through 30(±7) days after the last dose of study medication
  Ctrough of HY-0102 was observed directly from data.
Tmax (Time of maximum observed serum concentration) of HY-0102 | From first dose through 30(±7) days after the last dose of study medication
  Tmax of HY-0102 was observed directly from data as time of Cmax.
AUC(0-T) [Area under the concentration-time curve from time zero to the last quantifiable concentration] of HY-0102 | From first dose through 30(±7) days after the last dose of study medication
  AUClast of HY-0102 was determined by linear/log trapezoidal method.
AUC(tau) [Area under the concentration-time curve in one dosing interval] of HY-0102 | From first dose through 30(±7) days after the last dose of study medication
  AUCtau of HY-0102 was determined using linear/log trapezoidal method.
AUC(inf) [Area under the concentration-time curve from time zero to infinity and the extrapolated area] of HY-0102 | From first dose through 30(±7) days after the last dose of study medication
  AUCinf = AUClast + (Clast*/kel), where Clast* is the estimated concentration at the time of the last measurable concentration and kel is the terminal phase rate constant calculated as the absolute value of the slope of a linear regression during the terminal phase of the natural log-transformed concentration time profile.
T1/2 (Elimination half life) of HY-0102 | From first dose through 30 days (+/- 7 days) after the last dose of study medication
  T1/2 of HY-0102 was observed directly from data.
CL(Total body clearance) of HY-0102 | From first dose through 30(±7) days after the last dose of study medication
  CL = Dose/AUCinf for Cycle 1 and Dose/AUCtau for Cycle 2. It was reported in units of milliliter per hour per kilogram (mL/hr/kg).
Vss (Volume of distribution at steady state) of HY-0102 | From first dose through 30(±7) days after the last dose of study medication
  Vss = CL × MRT, where CL is clearance and MRT is the mean residence time after intravenous administration.
Anti-drug Antibody (ADA) and Neutralizing Antibody (NAb) | From first dose through 30(±7) days after the last dose of study medication
  To assess the immunogenicity of HY-0102
ORR (confirmed complete or partial response) | FU period/EOS visits every 3 months (± 14 days) after the EOT visit for 6 months
  According to the modified RECIST1.1 for immune based therapeutics (iRECIST) to assess anti-tumor activity of HY-0102.
DCR (confirmed response or stable disease lasting for at least 6 months) | FU period/EOS visits every 3 months (± 14 days) after the EOT visit for 6 months
  According to the modified RECIST1.1 for immune based therapeutics (iRECIST) to assess anti-tumor activity of HY-0102.
Duration of Response (DoR) | FU period/EOS visits every 3 months (± 14 days) after the EOT visit for 6 months
  According to the modified RECIST1.1 for immune based therapeutics (iRECIST) to assess anti-tumor activity of HY-0102.
Progression Free Survival (PFS) | FU period/EOS visits every 3 months (± 14 days) after the EOT visit for 6 months
  According to the modified RECIST1.1 for immune based therapeutics (iRECIST) to assess anti-tumor activity of HY-0102.
PD parameters: receptor occupancy (RO) of HY-0102 | From first dose through 30(±7) days after the last dose of study medication
  RO of HY-0102 of red blood cells, white blood cells, platelets and neoplastic cells in peripheral blood.

OTHER OUTCOMES:
Biomarkers | From first dose through 30(±7) days after the last dose of study medication
  Cytokine, NKG2A receptor, PBMC, HLA-E, TIL, cytokine, etc. This was an exploratory endpoint and no data were collected.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Sarah Cannon Research Institute, Orlando, Florida
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Texas Oncology, Tyler, Texas